CLINICAL TRIAL: NCT02038244
Title: Integrative Medicine for Chronic Pain - Process-Outcome-Study in the Context of an Internal Medicine Ward for Integrative Medicine
Brief Title: Integrative Medicine for Chronic Pain
Acronym: POSITIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Holger Cramer, Postdoctoral Researcher, Universität Duisburg-Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135393-BO
Record Dates: First submitted 2014-01-09; First posted 2014-01-16 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Integrative Medicine (Experimental)
  Interventions: Other: Multimodal integrative medicine inpatient treatment program

INTERVENTIONS:
Other: Multimodal integrative medicine inpatient treatment program

SUMMARY:
In this study, the effects of a 14-day inpatient treatment in an internal medicine ward for integrative medicine on pain, disability, quality of life, satisfaction with life, depression, and anxiety will be investigated. Furthermore the influence of potential process variables will be evaluated.

Effects will be measured after completion of the program (2 weeks), and at 6 months follow up after start of the program.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with any chronic pain condition
* at least 6 months pain duration
* written informed consent

Exclusion Criteria:

* participation in any other clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 14 days
  VAS

SECONDARY OUTCOMES:
Pain Intensity | 6 months
  VAS
Pain Disability | 14 days, 6 months
  - German Pain Questionnaire
Health-related quality of life | 14 days, 6 months
  Short Form (36) Health Survey
Life satisfaction | 14 days, 6 months
  Brief Multidimensional Life Satisfaction Scale
Depression | 14 days, 6 months
  Beck Depression Inventory
Acceptance | 14 days, 6 months
  Emotional/Rational Disease Acceptance Questionnaire
Mindfulness | 14 days, 6 months
  Conscious Presence and Self Control (CPSC) Scale
Subjective stress | 14 days, 6 months
  Perceived Stress Scale
Easiness of life | 14 days, 6 months
  Questionnaire on emotional and physical reactions
Ability and will to change | 14 days, 6 months
  Ability and will to change Questionnaire
Safety | 14 days, 6 months
  Adverse events
Pain Disability | 14 days, 6 months
  - Pain Disability Index

OTHER OUTCOMES:
Body awareness | 14 days, 6 months
  Translated body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Body Awareness Questionnaire (BAQ) (Shields 1989)
Body responsiveness | 14 days, 6 months
  Translated body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  * Body Responsiveness Scale (BRS)(Daubenmier 2005)
Body awareness and dissociation | 14 days, 6 months
  Translated body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Scale of Body Connection (SBC) (Price and Thompson 2007)
Postural awareness | 14 days, 6 months
  Newly developed body awareness questionnaire will be validated. It will further be used for mediation and moderator analysis with the outcomes.
  - Postural Awareness Scale (PAS) (Cramer et al.)
Body awareness | 14 days, 6 months
  The DKB will be used for mediation and moderator analysis with the outcomes and for validation purposes.
  - Dresden Body Image Questionnaire (DKB) (Pöhlmann et al., 2007)
Daily log | 2 weeks
  Daily rating of pain and well-being on a 100mm visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany